CLINICAL TRIAL: NCT05049915
Title: Evaluation of the Clinical Effectiveness of Bioactive Glass (S53P4) in the Treatment of Non-unions of the Tibia and Femur: a Randomized Controlled Non-inferiority Trial
Brief Title: Evaluation of the Clinical Effectiveness of Bioactive Glass (S53P4) in the Treatment of Tibia and Femur Non-unions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sebastian Findeisen (Other)
Collaborators: Bonalive Biomaterials Ltd (Industry)
Responsible Party: Sponsor-Investigator, Sebastian Findeisen, Intern, University Hospital Heidelberg
Organization: University Hospital Heidelberg (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-472/2017
Record Dates: First submitted 2021-06-08; First posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Pseudoarthrosis of Bone
MeSH Terms: interventions — Radioimmunoassay

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Masquelet technique: bioactive glass (Experimental)
  Interventions: Device: bioglass (S53P4)
- Masquelet technique: RIA + TCP (Active Comparator)
  Interventions: Device: RIA and TCP

INTERVENTIONS:
Device: bioglass (S53P4) — surgical procedure: Masquelet defect augmentation with bioglass
  Arms: Masquelet technique: bioactive glass
Device: RIA and TCP — surgical procedure: Masquelet defect augmentation with RIA and TCP
  Arms: Masquelet technique: RIA + TCP

SUMMARY:
Abstract Background: Treatment of non-union remains challenging and often necessitates augmentation of the resulting defect with an autologous bone graft (ABG). ABG is limited in quantity and its harvesting incurs an additional surgical intervention leaving the risk for associated complications and morbidities. Therefore, artificial bone graft substitutes that might replace autologous bone are needed. S53P4-type bioactive glass (BaG) is a promising material which might be used as bone graft substitute due to its osteostimulative, conductive and antimicrobial properties. In this study, the investigators plan to examine the clinical effectiveness of BaG as a bone graft substitute in Masquelet therapy in comparison with present standard Masquelet therapy using an ABG with tricalciumphosphate to fill the bone defect.

Methods/design: This randomized controlled, clinical non-inferiority trial will be carried out at the Department of Orthopedics and Traumatology at Heidelberg University. Patients who suffer from tibial or femoral non-unions with a segmental bone defect of 2-5 cm and who are receiving Masquelet treatment will be included in the study. The resulting bone defect will either be filled with autologous bone and tricalciumphosphate (control group, N = 25) or BaG (S53P4) (study group, N = 25). Subsequent to operative therapy, all patients will receive the same standardized follow-up procedures. The primary endpoint of the study is union achieved 1year after surgery.

Discussion: The results from the current study will help evaluate the clinical effectiveness of this promising biomaterial in non-union therapy. In addition, this randomized trial will help to identify potential benefits and limitations regarding the use of BaG in Masquelet therapy. Data from the study will increase the knowledge about BaG as a bone graft substitute as well as identify patients possibly benefiting from Masquelet therapy using BaG and those who are more likely to fail, thereby improving the quality of non-union treatment.

ELIGIBILITY:
Inclusion Criteria:

* pseudarthrosis of the tibia or femur
* bone defect < 5 cc
* surgical treatment with Masquelet technique

Exclusion Criteria:

* age under 18
* disagreement
* patients who require amputation of the affected limb

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of participants with osseus consolidation evaluation via x-ray | 1 year post-operative Masquelet step II
  x-ray in 2 planes; union = cortical bridging of at least three out of four cortices

SECONDARY OUTCOMES:
12-item Short Form Survey (SF-12) | 1 year post-operative Masquelet step II
  Quality of life: Physical Score 23.99938(lowest/worst)-56.57706(highest/best), Mental Score 19.06444(lowest/worst)-60.75781 (highest/best)
Perfusion | 3 months post-operative Masquelet step II
  Real-time microperfusion assessment using Contrast enhanced ultra-sound (CEUS), contrasting agent: SonoVue. Objective perfusion quantification (using VueBox). Evaluation of characteristic perfusion parameters such as: wash-in rate, wash-in perfusion index
Rate of participants with osseus consolidation evaluation via CT | 1 year post-operative Masquelet step II
  union = cortical bridging of at least three out of four cortices

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Schmidmaier, Prof. Dr., Study Director — HTRG
Locations (1):
- University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
anonymized/pseudonymized, data that underlies results in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: after conclusion and evaluation of the study
Access Criteria: public
URL: https://pubmed.ncbi.nlm.nih.gov/29843766/

REFERENCES:
- [Background] Einhorn TA. The cell and molecular biology of fracture healing. Clin Orthop Relat Res. 1998 Oct;(355 Suppl):S7-21. doi: 10.1097/00003086-199810001-00003. PMID 9917622
- [Background] Schmidmaier G, Moghaddam A. [Long Bone Nonunion]. Z Orthop Unfall. 2015 Dec;153(6):659-74; quiz 675-6. doi: 10.1055/s-0035-1558259. Epub 2015 Dec 15. German. PMID 26670151
- [Background] Hak DJ, Fitzpatrick D, Bishop JA, Marsh JL, Tilp S, Schnettler R, Simpson H, Alt V. Delayed union and nonunions: epidemiology, clinical issues, and financial aspects. Injury. 2014 Jun;45 Suppl 2:S3-7. doi: 10.1016/j.injury.2014.04.002. PMID 24857025
- [Background] Giannoudis PV, Einhorn TA, Marsh D. Fracture healing: the diamond concept. Injury. 2007 Sep;38 Suppl 4:S3-6. doi: 10.1016/s0020-1383(08)70003-2. PMID 18224731
- [Background] Romano CL, Logoluso N, Meani E, Romano D, De Vecchi E, Vassena C, Drago L. A comparative study of the use of bioactive glass S53P4 and antibiotic-loaded calcium-based bone substitutes in the treatment of chronic osteomyelitis: a retrospective comparative study. Bone Joint J. 2014 Jun;96-B(6):845-50. doi: 10.1302/0301-620X.96B6.33014. PMID 24891588
- [Background] Valimaki VV, Aro HT. Molecular basis for action of bioactive glasses as bone graft substitute. Scand J Surg. 2006;95(2):95-102. doi: 10.1177/145749690609500204. PMID 16821652
- [Background] Lindfors N, Geurts J, Drago L, Arts JJ, Juutilainen V, Hyvonen P, Suda AJ, Domenico A, Artiaco S, Alizadeh C, Brychcy A, Bialecki J, Romano CL. Antibacterial Bioactive Glass, S53P4, for Chronic Bone Infections - A Multinational Study. Adv Exp Med Biol. 2017;971:81-92. doi: 10.1007/5584_2016_156. PMID 28050878
- [Background] Lindfors NC, Hyvonen P, Nyyssonen M, Kirjavainen M, Kankare J, Gullichsen E, Salo J. Bioactive glass S53P4 as bone graft substitute in treatment of osteomyelitis. Bone. 2010 Aug;47(2):212-8. doi: 10.1016/j.bone.2010.05.030. PMID 20624692
- [Background] van Gestel NA, Geurts J, Hulsen DJ, van Rietbergen B, Hofmann S, Arts JJ. Clinical Applications of S53P4 Bioactive Glass in Bone Healing and Osteomyelitic Treatment: A Literature Review. Biomed Res Int. 2015;2015:684826. doi: 10.1155/2015/684826. Epub 2015 Oct 4. PMID 26504821
- [Background] Kokubo T, Takadama H. How useful is SBF in predicting in vivo bone bioactivity? Biomaterials. 2006 May;27(15):2907-15. doi: 10.1016/j.biomaterials.2006.01.017. Epub 2006 Jan 31. PMID 16448693
- [Background] Stoor P, Apajalahti S, Kontio R. Regeneration of Cystic Bone Cavities and Bone Defects With Bioactive Glass S53P4 in the Upper and Lower Jaws. J Craniofac Surg. 2017 Jul;28(5):1197-1205. doi: 10.1097/SCS.0000000000003649. PMID 28538076
- [Background] Stoor P, Pulkkinen J, Grenman R. Bioactive glass S53P4 in the filling of cavities in the mastoid cell area in surgery for chronic otitis media. Ann Otol Rhinol Laryngol. 2010 Jun;119(6):377-82. doi: 10.1177/000348941011900603. PMID 20583735
- [Background] Kankare J, Lindfors NC. Reconstruction of Vertebral Bone Defects using an Expandable Replacement Device and Bioactive Glass S53P4 in the Treatment of Vertebral Osteomyelitis: Three Patients and Three Pathogens. Scand J Surg. 2016 Dec;105(4):248-253. doi: 10.1177/1457496915626834. Epub 2016 Jun 23. PMID 26929284
- [Background] Fischer C, Frank M, Kunz P, Tanner M, Weber MA, Moghaddam A, Schmidmaier G, Hug A. Dynamic contrast-enhanced ultrasound (CEUS) after open and minimally invasive locked plating of proximal humerus fractures. Injury. 2016 Aug;47(8):1725-31. doi: 10.1016/j.injury.2016.05.005. Epub 2016 May 14. PMID 27242329
- [Background] Fischer C, Preuss EM, Tanner M, Bruckner T, Krix M, Amarteifio E, Miska M, Moghaddam-Alvandi A, Schmidmaier G, Weber MA. Dynamic Contrast-Enhanced Sonography and Dynamic Contrast-Enhanced Magnetic Resonance Imaging for Preoperative Diagnosis of Infected Nonunions. J Ultrasound Med. 2016 May;35(5):933-42. doi: 10.7863/ultra.15.06107. Epub 2016 Apr 1. PMID 27036169
- [Background] Fischer C, Nissen M, Schmidmaier G, Bruckner T, Kauczor HU, Weber MA. Dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) for the prediction of non-union consolidation. Injury. 2017 Feb;48(2):357-363. doi: 10.1016/j.injury.2017.01.021. Epub 2017 Jan 9. PMID 28088373
- [Background] Haubruck P, Kammerer A, Korff S, Apitz P, Xiao K, Buchler A, Biglari B, Zimmermann G, Daniel V, Schmidmaier G, Moghaddam A. The treatment of nonunions with application of BMP-7 increases the expression pattern for angiogenic and inflammable cytokines: a matched pair analysis. J Inflamm Res. 2016 Sep 22;9:155-165. doi: 10.2147/JIR.S110621. eCollection 2016. PMID 27703392
- [Background] Moghaddam A, Breier L, Haubruck P, Bender D, Biglari B, Wentzensen A, Zimmermann G. Non-unions treated with bone morphogenic protein 7: introducing the quantitative measurement of human serum cytokine levels as promising tool in evaluation of adjunct non-union therapy. J Inflamm (Lond). 2016 Jan 22;13:3. doi: 10.1186/s12950-016-0111-x. eCollection 2016. PMID 26807043
- [Background] Tanner MC, Heller R, Westhauser F, Miska M, Ferbert T, Fischer C, Gantz S, Schmidmaier G, Haubruck P. Evaluation of the clinical effectiveness of bioactive glass (S53P4) in the treatment of non-unions of the tibia and femur: study protocol of a randomized controlled non-inferiority trial. Trials. 2018 May 30;19(1):299. doi: 10.1186/s13063-018-2681-9. PMID 29843766

DOCUMENTS (1):
  • Study Protocol (2017-08-16): https://cdn.clinicaltrials.gov/large-docs/15/NCT05049915/Prot_000.pdf